CLINICAL TRIAL: NCT01035580
Title: Phase I Trial on Safety and Pharmacokinetics of Intravaginal Curcumin in Normal Female Subjects
Brief Title: Trial on Safety and Pharmacokinetics of Intravaginal Curcumin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lisa Flowers, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00020139
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Uterine Cervical Dysplasia
Keywords: chemoprevention; curcumin; pharmacokinetics; safety
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- curcurim (Experimental): This was a 3 + 3 dose escalation trial starting at 500 mg of cur cumin capsules administered daily intravaginally for 14 days. The dose increased after safety was demonstrated in 3 subjects by 500 mg up to a max of 2000 mgs.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Curcumin 500 mg capsules will be inserted intravaginally once daily for 14 days for a maximum daily dosage of 2000 mg
Drug: curcumin — all patients received the drug
  Other Names: Sabinsa Curcumin Capsules

SUMMARY:
The main objective of this study is to determine the maximum tolerable dose and safety of intravaginal curcumin in a normal population of women (women with no evidence of cervical cytological abnormalities by pap testing).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45 years of age at enrollment
* Currently using a reliable birth control method (oral contraceptive pills, DepoProvera or permanent sterilization)
* Able to provide written informed consent
* Provide male partner notification letter
* Have a Pap test negative pap (no cervical intraepithelial lesions) within 45 days prior to screening
* Have regular monthly menses (every 21-35 days) or amenorrhea due to hormonal contraceptive use
* Agree to undergo pelvic exam and colposcopy per protocol
* Able and willing to complete Study Diary
* Agree to wear condoms during all acts of vaginal intercourse or abstain from vaginal intercourse during the 14 days
* Agree to abstain from sexual intercourse for 48 hours prior to the enrollment visit
* Agree to insert curcumin gelatin capsules as required per protocol
* Agree to abstain from nonsteroidal anti-inflammatory drugs (NSAIDS) during the 14 days
* Agree to abstain from all products containing curcumin or food consumption of curcumin during the 14 days
* Agree to abstain from the following activities for at least 48 hours prior to enrollment through the Day 14 visit:insertion of objects into the vagina except for a penis, receiving oral or anal sex,using a diaphragm, cervical cap, female condom, or vaginal contraceptive ring,using vaginal products other than the study gelatin capsules, including douches, lubricants, spermicide or feminine hygiene products,participating in other vaginal cream or contraceptive studies
* Agree to testing for HIV status via enzyme immunoassay (EIA)/Western Blot

Exclusion Criteria:

* Are post-menopausal
* Have had a hysterectomy with removal of the cervix
* Have a clinically significant chronic medical condition that is considered progressive, including: coronary disease, congestive heart failure, chronic obstructive lung disease, diabetes mellitus, chronic renal disease, active peptic ulcer disease, chronic hepatic disease, multiple sclerosis, seizure disorder requiring medication, and a coagulation or platelet disorder. Chronic nonprogressive or intermittent syndromes are not excluded, including migraine headaches, mild reactive airways disease, controlled hypertension, stable pain syndromes, or benign gastric reflux.
* Have an intrauterine device (IUD) as a form of birth control
* Have any history of malignancy or current (within 45 days of screening) pap with cervical intraepithelial lesions.
* Currently has documented lacerations on visual inspection present on the cervix, vagina, vulva or perineum.
* Are pregnant or planning to become pregnant in the next three months
* Are currently breastfeeding
* Have a history of sensitivity or allergy to any compound used in this study
* Have Grade 2 or higher renal or hematologic abnormality, as defined by the Table for Grading the Severity of Adult Adverse Events or at screening have a positive bacterial urine culture. Women with a positive bacterial urine culture at screening will be allowed to enroll after appropriate treatment if repeat evaluation is normal.
* In the three months prior to enrollment have had any of the following:Treatment for Cervical disease or any other gynecologic surgery,A pregnancy or an abortion, An IUD,Breakthrough menstrual bleeding or vaginal bleeding during or following vaginal intercourse
* Signs, as seen on pelvic exam at screening, consistent with an STD including vaginitis, cervicitis or genital ulcers
* Signs, as seen on pelvic exam, of genital trauma
* Signs of genital tract infection from laboratory evaluations. Women with Candida vaginitis or bacterial vaginosis at screening will be allowed to enroll after appropriate treatment and if repeat evaluation is normal.
* In the three months prior to enrollment have had any of the following:History of treatment for or a diagnosis with a new STD,Genital herpes simplex virus infection or outbreak,Exchanged sex for money, drugs or gifts
* Are currently using, or in the last year have used intravenous drugs (except for therapeutic use), cocaine or other recreational drugs, abused alcohol defined as alcohol use that has required hospital admission for detoxification and therapy.
* Have any other condition that in the opinion of the investigator might interfere with the evaluation of the study objectives.
* HIV positive

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to reach the maximum selected dose (MSD) or maximum tolerated dose (MTD) of intravaginal curcumin among Pap test negative women without causing a dose-limiting toxicity. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, Medical, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States